CLINICAL TRIAL: NCT03170440
Title: Non-invasive Vagal Nerve Stimulation and Sleep
Brief Title: Non-invasive Nerve Stimulation for PTSD and Sleep
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); North Florida/South Georgia Veterans Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB201700541; i01 rx003140-01a (Other Grant/Funding Number: Department of Veterans Affairs); I01RX003140-01 (NIH)
Record Dates: First submitted 2017-05-23; First posted 2017-05-31 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Post Traumatic Stress Disorder; Traumatic Brain Injury
Keywords: Nerve stimulation; sleep deprivation
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic; Sleep Deprivation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Noninvasive nerve stimulation type I (Experimental): This group will receive one type of nerve stimulation
  Interventions: Device: Transcutaneous nerve stimulation location 1
- Noninvasive nerve stimulation type II (Active Comparator): This group will receive second type of nerve stimulation
  Interventions: Device: Transcutaneous nerve stimulation location 1

INTERVENTIONS:
Device: Transcutaneous nerve stimulation location 1 — Non-invasive stimulation by transcutaneous electrical nerve stimulation device in test location

SUMMARY:
In this study, our objective is to determine the effect of two different nerve stimulation types in changing sleep architecture.

DETAILED DESCRIPTION:
Persons suffering from PTSD or mild TBI may suffer from sleep deprivation. The purpose of this study is to explore options to improve sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* veterans with history of PTSD with and without history of mild TBI

Exclusion Criteria with:

* history of severe psychiatric illness unrelated to PTSD or TBI
* other medical conditions of severity that may impair cognition
* current illicit or prescription drug abuse
* breathing disorder requiring constant use of oxygen

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 221 (Estimated)
Dates: Start 2017-11-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
Physiological sleep architectural quality | up to 8 hours
  Polysomnography

CONTACTS AND LOCATIONS:
Overall Officials: John Williamson, Ph.D., Principal Investigator — University of Florida
Locations (3):
- United States (3):
  - UF Health Jacksonville, Gainesville, Florida
  - University of Florida, Gainesville, Florida
  - UF Health Jacksonville, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: No